CLINICAL TRIAL: NCT05031455
Title: Mechanisms of Dupilumab in AERD - Effects on Aspirin Hypersensitivity Response, With a Focus on Innate Type 2 Inflammatory Responses
Brief Title: Mechanisms of Dupilumab in AERD
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Scripps Clinic (Other)
Collaborators: University of California, San Diego (Other); Regeneron Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Andrew White, Director, Aspirin Exacerbated Respiratory Disease Clinic, Scripps Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHUCSD06242020
Record Dates: First submitted 2021-08-19; First posted 2021-09-02 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-04

CONDITIONS: Aspirin-exacerbated Respiratory Disease
MeSH Terms: interventions — dupilumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Aspirin Challenge (Experimental): All subjects will undergo a standardized aspirin challenge
  Interventions: Drug: Aspirin Challenge

INTERVENTIONS:
Drug: Aspirin Challenge — Dupilumab is a fully human monoclonal antibody that blocks the receptor component for IL-4 and IL-13, which are key drivers of type 2 inflammation. All subjects will be prescribed this at standard 300mg subcutaneous dosing every 2 weeks. The intervention will be the response to aspirin challenge.
  All 16 subjects will receive dupilumab. All subjects will undergo an aspirin challenge/desensitization procedure. It is estimated that 50% of subjects will have a respiratory reaction to aspirin and 50% will not. There will not be any randomization.
  Other Names: Dupixent

SUMMARY:
Aspirin-Exacerbated Respiratory Disease (AERD), although uncommon in the general population, is an important phenotype of severe asthma and nasal polyposis where it occurs in 15% of severe asthmatics, and up to 30% of those with nasal polyposis. An important therapy for AERD is aspirin therapy after desensitization (ADAT). This is an inexpensive and proven therapy to improve the burden of sinus disease in AERD. Aspirin desensitization is the mechanism by which tolerance is induced in AERD patients. This is a 1-2 day outpatient procedure whereby increasing doses of aspirin are administered and the patients invariably experience some degree of hypersensitivity reactions.

It is important to understand the effect of medications on the aspirin desensitization. It is known that the leukotriene modifier medications decrease the severity of the reactions in AERD. Other treatments such as antihistamines and the biologic agent omalizumab might have an effect on either blocking or blunting reactivity in AERD during desensitization.

Dupilumab is a new respiratory biologic approved for atopic dermatitis, eosinophilic asthma and nasal polyposis. As such, it is well situated to be used for many AERD patients whose disease cannot be well controlled. The effect of dupilumab on the aspirin desensitization process and reaction is unknown and is the topic of this investigation.

The primary objective is to determine the effect of dupilumab on reactions during aspirin challenge/desensitization.

ELIGIBILITY:
Inclusion Criteria:

* Subjects >18 years old with Aspirin-Exacerbated Respiratory Disease

This is diagnosed via either a positive oral aspirin or intranasal ketorolac challenge OR a history of at least two stereotypical hypersensitivity reactions to aspirin leading to nasal-ocular symptom and/or asthmatic symptoms.

* Current treatment with dupilumab at standard asthma/nasal polyposis dosing of 300mg subcutaneously every 2 weeks for a minimum of 12 weeks.
* All subjects will be required to have a known history of nasal polyposis either via imaging, endoscopy, or nasal examination

Exclusion Criteria:

* History of gastrointestinal reactions (severe abdominal pain with or without vomiting) during NSAID triggered events
* Unstable asthma or history of severe reactions during previous desensitization attempts
* inability to take montelukast pretreatment
* history of gastrointestinal bleeding or bleeding disorder
* pregnancy
* previous use of any other respiratory biologic in the past 3 months (omalizumab, tezepelumab, mepolizumab, reslizumab, benralizumab)
* need for systemic corticosteroids to stabilize asthma prior to challenge
* time from sinus surgery <1 month.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2024-03-25 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Rate of positive challenges to aspirin challenge | Aspirin challenge = 6 weeks after starting dupilumab/placebo. Aspirin challenge day = up to 8 hours
  Aspirin challenge reactions will be defined as either 1) >15% drop in FEV1 or 2) >25% drop in peak nasal inspiratory flow (PNIF) or 3) >5 point change in composite symptom score.
  Spirometry is a standardized measure of airflow obstruction used to define lower airway reaction to aspirin in AERD.
  Nasal inspiratory flow rates are measured using an inverted peak flow meter and have been correlated with nasal obstruction occurring during nasal reactions to aspirin in AERD.
  Symptom Score - symptoms are a typical part of an aspirin reaction with increase in congestion, itching, cough, and chest tightness.

CONTACTS AND LOCATIONS:
Locations (1):
- Scripps Clini, San Diego, California, United States